CLINICAL TRIAL: NCT04729088
Title: Phase I Clinical Trial to Evaluate the Pharmacokinetic Profile of a Formulation With Isosorbide Mononitrate 0.5% Gel - Manufactured by Sanus Pharmaceutical Ltda, to Intra Anal Application in Healthy Males and Females' Subjects
Brief Title: Pharmacokinetics Trial of Isosorbide Mononitrate 0.5% Gel for Intra Anal Application in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor will no longer develop the experimental drug.
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAEP 56.003.19PC
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pharmacokinetics; Healthy Subjects
Keywords: Isosorbide Mononitrate; Pharmacokinetics; Intra anal application; Anal Fissure; Healthy volunteers
MeSH Terms: conditions — Fissure in Ano | interventions — isosorbide-5-mononitrate

STUDY DESIGN:
Intervention Model Description: Phase I, single-center, single-dose clinical trial (test drug), in which participants will receive the test drug intra-anal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Drug (Experimental): Isosorbide 0.5% gel
  Interventions: Drug: Isosorbide mononitrate

INTERVENTIONS:
Drug: Isosorbide mononitrate — Intra-anal application performed by the study physician of 2 g of the study drug

SUMMARY:
This is a Phase I trial to evaluate pharmacokinetics and safety of Isosorbide Mononitrate gel for intra anal administration in healthy subjects.

DETAILED DESCRIPTION:
This is a Phase I trial to evaluate the pharmacokinetics and safety of Isosorbide Mononitrate gel for intra anal administration. For the current study 2g of a 0,5% gel will be used (as part of a safety investigational profile with doses up to 2% in other studies).

The investigational product will be administered to the participants by the study physician as a single dose. Blood samples will be collected prior dose and up to 36:00 hours to characterize the pharmacokinetic profile.

Safety parameters, including adverse events, will be monitored by the study team during confinement (up to 24 hours post dose), at the 36 hour sample collection (ambulatory basis) and as reported by the subjects or verified at the discharge visit, up to 15 days after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged from 18 to 50 years-old;
* Good health conditions or without significant diseases, according to medical judgement, according to protocol requirements and study evaluations: medical history, blood pressure and heart rate measurements, physical examination, electrocardiogram (ECG) and screening laboratory test;
* Ability to understand the nature and objectives of the trial, including risks and adverse events;
* Willingness to proceed according to all study requirements, which shall be confirmed by Informed Consent Form signature;
* Agree to use safe contraceptive method.

Exclusion Criteria:

* Known to have hypersensitivity reaction to the studied drug or to chemically related compounds;
* History or presence of chronic gastrointestinal diseases or other condition that may interfere with drug absorption, distribution, metabolism or excretion;
* Maintenance therapy with any drug known to interact with the investigational drug, except contraceptives;
* History of liver, kidney, lung, gastrointestinal, epileptic, haematological or psychiatric disease; hypertension of any etiology; history of myocardial infarction, angina and / or heart failure or malignant neoplasms. Have any current disease, acute or chronic, in follow-up or treatment;
* Have active orificial pathology, such as hemorrhoidal thrombosis, acute or chronic anal fissures, as assessed by the study physician within 15 days from confinement;
* Electrocardiographic findings not recommended at the physician's discretion to participate in the study;
* History of cardiac (any), renal (renal exeresis or agenesis), gastrointestinal (partial or total removal of the esophagus, stomach, duodenum, jejunum, ileum, ascending colon, transverse colon, descending colon, sigmoid or rectum), liver or pancreas surgery;
* Screening laboratory test results outside normal ranges set by the clinical analysis laboratory, unless considered non-clinically significant by the Principal Investigator / Physician;
* Smoker (more than five cigarettes / day);
* Eating foods containing xanthine, including more than five cups of coffee or tea per day;
* Unusual eating habits, eg vegetarians;
* History of excessive alcohol consumption (drinking 4 or more alcoholic beverages in one day or 8 or more alcoholic beverages per week for women and 5 or more alcoholic beverages in one day or 15 or more alcoholic beverages per week for men);
* History of drug use;
* Use of regular medication within two weeks prior to initiation of treatment and the date of pre-confinement clinical assessment;
* Use of medication containing sildenafil, vardenafil or riociguate, up to 03 days before confinement;
* Use medication containing tadalafil up to 08 days before confinement;
* Use of any medication, except contraceptives or cases where, based on the half-life of the drug and / or active metabolites, complete elimination may be assumed;
* Hospitalization due to any reason up to eight weeks before the start of the trial treatment;
* Treatment with any drug known to have well established toxic potential in the large organs, within three months prior to the study;
* Participation in any other experimental research or administration of any experimental drug within six months prior to the commencement of this trial;
* Pregnancy or breastfeeding or wish to become pregnant during the trial period;
* Donation or loss of 450 mL or more of blood within the three months prior to the trial or donation of more than 1500 mL within the twelve months preceding the trial;
* Any condition that, according to the investigator's best judgement, precludes participation in this trial;
* Inability to lie down, preferably on the side, for 1 hour or as long as necessary at the doctor's discretion;
* Positive test for pregnancy;
* Breathalyzer test result greater than zero;
* Positive result for drug of abuse testing;
* Unavailability for registration on the National Register for Bioequivalence Studies (CNVB)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve from time zero to last (AUC 0-last) | 36 hours
Area under the plasma concentration versus time curve from time zero to infinite (AUC 0-inf) | 36 hours
Maximum (peak) plasma concentration (Cmax) | 36 hours
Time to reach maximum (peak) plasma concentration (Tmax) | 36 hours
  Time frame from drug administration to sampling time of maximum plasma concentration
Elimination rate constant (Ke) | 36 hours
Half life (t1/2) | 36 hours

SECONDARY OUTCOMES:
Number of adverse events | 15 days
Blood Pressure | 1 day
  Blood pressure (Systolic and Diastolic Blood Pressure) pre-dose, at each hour until 12 hours after dose and 24 hours after dose
Pulse | 1 day
  Pulse pre-dose, at each hour until 12 hours after dose and 24 hours after dose

CONTACTS AND LOCATIONS:
Overall Officials: José Pedrazzoli Jr., MD, Principal Investigator — CAEP - Centro Avançado de Estudos e Pesquisas Ltda.